CLINICAL TRIAL: NCT03990454
Title: A Phase 1, Open-label, Dose-escalationStudy of the Safety and Pharmacokinetics of the AXL Inhibitor SLC-391 Administered Orally to Subjects With Solid Tumours
Brief Title: Safety Study of SLC-391 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SignalChem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SLC-391-101
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor
Keywords: AXL Inhibitor; Solid Tumor

STUDY DESIGN:
Intervention Model Description: The study will employ a 3+3 dose-escalation design. Cohorts (same dose level) of 3 to 6 evaluable subjects will participate in a dose-escalation scheme in which the dose of SLC-391 will be increased in each consecutive cohort. Evaluation of a cohort of ≥ 3 subjects that have completed a 21-day cycle (cycle 1) is required prior to defining a new SLC-391 dose and schedule for the next cohort. Dose-escalation decisions by the Data Review Committee will take into account all available data including PK/pharmacodynamic data and the safety profile of prior cohorts. Based on all available emerging data, alternative dosing schedules, frequency, or dose reductions may be considered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): The starting dose will be 25 mg/day and subsequent doses will be determined after an internal review by Data Review Committee of all available safety, PK and PD data from the minimum required number of subjects who complete cycle 1. All dose-escalation decisions and the rationale for progressing to the next cohort will be documented.
  A subject may continue treatment with SLC-391 in 21-day cycles until the treatment discontinuation criteria are met.
  Interventions: Drug: SLC-391

INTERVENTIONS:
Drug: SLC-391 — SLC-391 is an AXL inhibitor

SUMMARY:
SLC-391 is a novel, potent and specific small molecule inhibitor of receptor tyrosine kinase AXL with desirable potency and pharmaceutical properties. It has demonstrated antiproliferative activity against different tumour cell lines in vitro and efficacy in different animal models including nonsmall cell lung cancer (NSCLC), chronic myeloid leukemia (CML) and (acute myeloid leukemia (AML) models. It has also exhibited strong synergy with other approved targeted therapies in different animal models.

This is the first clinical study with SLC-391. The goals of this study are to evaluate the safety, pharmacokinetic (PK), and pharmacodynamic profile of SLC-391, and then to identify a safe and pharmacologically active dose for evaluation in subsequent cohorts or clinical studies. In addition, change from baseline of possible blood biomarkers (soluble AXL and Gas 6) may be evaluated.

This is an open-label, multicentre, phase 1, dose-escalation, first in human study to evaluate the safety of SLC-391 administered orally (once or twice daily) in 21-day cycles to subjects with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older at the time of signing the informed consent.
* Have a histologically or cytologically confirmed diagnosis of a solid tumour malignancy that is advanced and/or metastatic or unresectable and for which standard or curative measures do not exist or are no longer effective.
* Have measurable disease as per the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 or as per a modified RECIST, if applicable.
* Have a performance status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Be able to ingest oral medication.
* Have adequate organ function,
* Have recovered to ≤ grade 1 from the effects of any prior cancer therapy, except for alopecia; irreversible neuropathy should have recovered to ≤ grade 2. Toxic effects also include laboratory test abnormalities.
* Be afebrile at baseline prior to SLC-391 administration (ie, < 38.0 °C).
* Have a life expectancy greater than 3 months, in the Investigator's opinion.
* The following time must have elapsed between previous therapy for cancer and first dose of SLC-391:

  1. At least 4 weeks since previous cancer-directed therapy, including investigational agents or devices (cytotoxic agents, targeted therapy including monoclonal antibodies, immunotherapy, hormonal therapy, and prior radiotherapy) with the exception of nitrosoureas/mitomycin where 6 weeks since these therapies.
  2. At least 4 weeks or 5 times the elimination half-life (whichever is shortest) of any investigational agents, including drugs, biologics, or combination products.
  3. At least 4 weeks since any major surgery.
* Sexually active women of child-bearing potential and sexually active male subjects with a female partner of child-bearing potential or pregnant must agree to use acceptable methods of contraception to avoid pregnancy from screening, for the duration of the study, and for 3 months after the last dose of study drug. Male subjects must also agree to refrain from donating sperm for the duration of the study, including during dose interruptions and for 3 months after the last dose administered.
* Be able and willing to provide signed informed consent and comply with the requirements, assessment schedule, dosing schedule, and restrictions listed in the informed consent form (ICF) and study protocol.

Exclusion Criteria:

* Prior use of any AXL inhibitor
* Localised or metastatic prostate cancer subjects who are concurrently receiving abiraterone or enzalutamide. Those subjects on stable (>3 months) anti-cancer hormonal therapy are allowed.
* Refractory nausea and vomiting, chronic gastrointestinal (GI) diseases, GI bleeding, ulceration, or perforation within 12 weeks prior to the first dose of the study drug, or significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of the study drug.
* History of myocardial infarction, unstable angina, congestive heart failure (New York Heart Association class ≥ III/IV), cerebrovascular accident, transient ischaemic attack, limb claudication at rest, stroke or subarachnoid hemorrhage, coagulopathy, deep vein thrombosis, pulmonary embolism in the 3 months prior to consent.
* Uncontrolled hypertension (≥ 160/100 mmHg).
* History of or ongoing symptomatic dysrhythmias, uncontrolled atrial or ventricular arrhythmias, or heart block (excluding 1st degree block, consisting of PR interval prolongation only). Controlled atrial fibrillation is allowed.
* QTcF interval > 480 msec.
* Severe respiratory illness that significantly impacts functional status in daily life including a known history of active tuberculosis (Mycobacterium tuberculosis).
* History of significant weight loss (≥ 7 kgs/15 lbs) within 4 weeks prior to the first dose of study drug.
* History of primary immunodeficiency or those with known human immunodeficiency virus (HIV), or known active hepatitis B (HBV; including core antibody and surface antigen; AntiHBc and HBsAg, respectively) or hepatitis C (HCV) infection. Note: No testing for HIV, Hepatitis B or C is required unless mandated by a local health authority.
* Active uncontrolled infection, or an unstable or severe intercurrent medical condition that requires treatment.
* History of solid organ transplant or bone marrow transplant.
* Any condition or illness that, in the opinion of the Investigator, would compromise subject safety or interfere with the evaluation of the safety of the study drug and jeopardises compliance with the protocol and study visits.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* History of prior malignancy, except for the following: curatively treated basal or squamous cell carcinoma of the skin (nonmelanoma skin cancer); cervical or vaginal intra-epithelial neoplasia; or noninvasive breast cancer in situ at screening. Subjects with other curatively treated malignancies who have had no evidence of metastatic disease and a > 2-year disease-free interval may be enrolled after approval by the Medical Monitor or SignalChem Lifesciences (SLC) designee.
* Females who are pregnant, planning to become pregnant, or breastfeeding.
* Hypersensitivity to the study drug or excipients (lactose, microcrystalline cellulose, magnesium stearate, and gelatin capsule shell).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as assessed by NCI-CTCAE v5.0 | 2 years
  To assess AEs as criteria of safety of oral SLC-391
Maximum Tolerated Dose of SLC-391 | 21 days
  To determine the maximum tolerated dose (MTD) of SLC-391

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SLC-391 | Day 1 predose through to Day 21 post-final dose
  Changes in AUC over time in subjects taking SLC-391 once or twice daily.
Maximum Observed Plasma Concentration (Cmax) | Day 1 predose through to Day 21 post-final dose
  Cmax is the maximum observed plasma concentration in ng/mL
Time to the Maximum Observed Plasma Concentration (Tmax) | Day 1 predose through to Day 21 post-final dose
  Tmax is the time in hours to reach Cmax following dosing
Terminal elimination half-life (t1/2) | Day 1 predose through to Day 21 post-final dose
  The time in hours required for the plasma level of the study drug to decrease by one-half during the terminal elimination phase
Recommended Dose of SLC-391 for future trials | 2 years
  Determine the recommended phase 2 dose (RP2D) of SLC-391
Preliminary efficacy of SLC-391 | 2 years
  Determine tumour response defined by the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 to SLC-391
Number of Participants with Clinically Significant Changes From Baseline in Laboratory Parameters | 2 years
  Laboratory investigation includes hematology, biochemistry, urinalysis, and Serology.
Number of Participants with Clinically Significant Changes From Baseline in Vital Signs | 2 years
  Vital sign measurements includes blood pressure, heart rate, respiratory temperature, and oral temperature.
Number of Participants with Clinically Significant Changes From Baseline in electrocardiogram (ECGs) Findings | 2 years
  ECG parameters includes heart rate, PR interval, QRS, QT, and QTcF.
Number of Participants with Clinically Significant Changes From Baseline in physical examinations | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zaihui Zhang, PhD, Study Director — SignalChem Lifesciences Corporation
Locations (3):
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No